CLINICAL TRIAL: NCT00119561
Title: Testing the Effectiveness of Telephone Support for Dementia Caregivers
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 03-287
Record Dates: First submitted 2005-07-05; First posted 2005-07-13 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2014-07

CONDITIONS: Dementia; Alzheimer Disease
Keywords: Caregiver; Dementia; Alzheimer Disease; Telephone; Randomized Controlled Trials
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Telephone support groups
  Interventions: Behavioral: Telephone Support
- Arm 2 (No Intervention): Usual VA care

INTERVENTIONS:
Behavioral: Telephone Support — Each telephone support group of 5 caregivers and a group leader met 14 times over a year. The hour calls were semi-structured with an educational component and a support component, led by a trained Group Leader. Topics included knowledge of dementia, safety, caregiver health and well being, communication, managing behavioral challenges and caregiver stress and coping.
  Arms: Arm 1

SUMMARY:
The primary goal of the study is documentation of effectiveness of telephone support groups to reduce caregiver burden and stress. Caregivers who participate in intervention (Telephone Support) should experience lower levels of stress, burden and health care utilization (lower use of psychotropic drugs, fewer scheduled/unscheduled medical visits, lower rates of institutionalization, more efficient use of time in managing care recipient problems) compared to those caregivers in Usual Care.

DETAILED DESCRIPTION:
Background: Caregiving can severely limit caregivers' lives. In order to keep their family member at home, dementia caregivers often experience physical and psychological strain, social isolation, loss of time for self, and inability to obtain and/or afford assistance with caregiving tasks. The amount of time spent in providing care for a family member with dementia contributes to these problems. Dementia caregivers report spending around 18 hours per day in caregiving tasks and 3 hours per day in supervision. The high levels of stress involved in caring for a dementia patient and the widespread lack of training in such care can lead to a vicious cycle of ever-increasing health care dependency, first for the patient and secondly for informal caregivers. Telephone Support Groups have the potential to address caregivers' stress, isolation and education about dementia and its management, leading to sustainable informal caregiving and lower healthcare use and overall VHA expenditures for the veteran patient with dementia.

Objectives: Study objectives are to 1) examine Telephone Support Groups' effectiveness for caregivers, 2) determine whether Telephone Support results in decreases in VHA health care use and costs for the veteran, and decreased VHA and/or non-VHA use and costs for the caregiver, and 3) examine the intervention's effect on caregivers' time spent providing care. The long-term objective is to develop and disseminate the protocol and materials for effective Telephone Support Groups that can be used across the VHA system.

Methods: This randomized clinical trial of 154 caregivers (Black/African American, White/Caucasian, rural, urban) compared dementia caregivers participating in Telephone Support Groups to caregivers whose family members with dementia were receiving usual care. Either the caregiver or the patient had to be a veteran receiving care at the VAMC Memphis. In the treatment condition, there were 15 year-long support groups of one trained group leader and 5 to 6 caregivers. Each support group met 14 times. The one hour calls were semi-structured conference calls with education, coping skills and cognitive restructuring, and support components. A Caregiver Notebook with information on each topic provided materials for the educational sessions. Topics included knowledge of dementia, safety, caregiver health and well being, communication, managing behavioral challenges, and caregiver stress and coping. A workshop focusing on the same behavior management and stress topics was offered to Usual Care caregivers at the end of their participation.

Data were collected in caregivers' homes by trained Research Associates at baseline, six and twelve months. VHA health care use and data for the veteran were based on the Patient Treatment File (PTF) and the Outpatient Clinic File (OPC) and costs data used the Health Economics Resource Center (HERC) Average Cost Data Sets.

ELIGIBILITY:
Inclusion Criteria:

Caregiver

* Age: 21 years or older
* Family member of the care recipient
* Must live with care recipient or share cooking facilities
* Must have a telephone
* Must plan to remain in the area for the duration of the intervention and follow-up
* Caregiver role for more than 6 months
* Must provide an average of 4 hours of supervision or direct assistance per day for the care recipient
* Risk Screening Tool: must have a total score of at least 1 for question 36, and a total of at least 2 for questions 38-40 (on the Screening Form)

Care Recipient

* NINCDS (MD diagnosis) or cognitive impairment (raw score on MMSE of 23 or less)
* Must be a Veteran with dementia or being cared for by a Veteran who receives services at the Memphis VAMC

Exclusion Criteria:

Caregiver

* Active treatment (chemotherapy; radiation therapy) for cancer
* Imminent placement of care recipient into a nursing home (within 6 months)
* SPMSQ: > 4 errors

Care Recipient

* History of Parkinson's Disease or a stroke with no reported decline in memory over the past year
* Active treatment (chemotherapy or radiation therapy) for cancer
* More than three acute medical hospitalizations in the past year (other than psychiatric or Alzheimer's Disease related admissions)
* Schizophrenia (onset of delusions before age 45) or other severe mental illness
* Dementia secondary to head trauma (probable)
* Blindness or deafness if either disability prohibits them from data collection or participation in the interventions
* MMSE = 0 and Bedbound (routinely confined to bed or chair for at least 22 hours a day, for at least 4 of the last 7 days)
* Planned nursing home admission in 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2005-02; Primary Completion 2007-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
General well-being (revised Rand General Well-Being Scale); and caregiver's level of distress with care recipient behaviors (Revised Memory and Behavior Problems Checklist). Data is collected at baseline, 6 and 12 months in a face to face interview. | 6 and 12 months

SECONDARY OUTCOMES:
Cost-Effectiveness | 6 and 12 months
Time spent providing care | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Linda Olivia Nichols, PhD, Principal Investigator — Memphis VA Medical Center, Memphis, TN
Locations (1):
- Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee, United States

REFERENCES:
- [Result] Nichols LO, Martindale-Adams JL, Burns R, Graney MJ, Zuber JK, Kennedy SE. Potential explanations for control group benefit. Clin Trials. 2012 Oct;9(5):588-95. doi: 10.1177/1740774512455876. Epub 2012 Aug 23. PMID 22917945
- [Result] Martindale-Adams J, Nichols LO, Burns R, Graney MJ, Zuber J. A trial of dementia caregiver telephone support. Can J Nurs Res. 2013 Dec;45(4):30-48. doi: 10.1177/084456211304500404. PMID 24617278